CLINICAL TRIAL: NCT00053924
Title: A Phase 2 Study Of Perifosine As Second Line Therapy For Advanced Pancreatic Carcinoma
Brief Title: Perifosine in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-015; CDR0000269586 (Registry Identifier: PDQ (Physician Data Query)); NCI-5983
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage II pancreatic cancer; adenocarcinoma of the pancreas; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — perifosine

INTERVENTIONS:
Drug: perifosine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of perifosine in treating patients who have locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of perifosine, in terms of 6-month survival, in patients with advanced adenocarcinoma of the pancreas.
* Determine the safety and tolerability of this drug in these patients.
* Determine median survival time and the 1-year survival rate of patients treated with this drug.
* Determine the objective response rate (partial and complete), response duration, and time to progression in patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: Patients receive oral perifosine daily for 3 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 17-37 patients will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas not amenable to curative local therapy

  * Metastatic OR locally advanced
* No known brain metastases
* No ascites that required therapeutic paracentesis on at least 2 occasions within the past 6 weeks

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN (5 times ULN with liver metastases)

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Gastrointestinal

* No gastrointestinal (GI) tract disease resulting in the inability to take oral medication or a requirement for IV alimentation
* No uncontrolled inflammatory bowel disease
* No active peptic ulcer disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to perifosine
* No other active malignant disease that could interfere with interpretation of study results
* No ongoing active infection
* No other uncontrolled concurrent illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 1 prior chemotherapy regimen for metastatic or locally advanced disease

  * Prior chemotherapy, given as a radiosensitizer, allowed in addition to single-line therapy
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* Not specified

Radiotherapy

* At least 3 weeks since prior radiotherapy likely to have myelotoxic effects (more than 3,000 cGy to fields including substantial marrow) and recovered

Surgery

* No prior GI surgery affecting absorption

Other

* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05; Primary Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J. Moore, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (3):
- Canada (3):
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario